CLINICAL TRIAL: NCT01340677
Title: An Open-Label, Single-Dose, Randomized, 3-Period, Crossover Study to Evaluate the Pharmacokinetic Dose Proportionality of Canagliflozin of 50, 100, and 300 mg Under Fasted Conditions in Healthy Subjects
Brief Title: A Pharmacokinetic Dose Proportionality Study of Canagliflozin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Director, Clinical Pharmacology, Johnson & Johnson Pharmaceutical Research and Development, L.L.C.
Model: Crossover | Masking: None
Other Study IDs: CR018277; 28431754DIA1015; 2010-023251-28
Record Dates: First submitted 2011-04-21; First posted 2011-04-22 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Healthy
Keywords: Canagliflozin (JNJ-28431754); Pharmacokinetic; Dose proportionality
MeSH Terms: interventions — Canagliflozin

ARMS (1):
- 001 (Experimental): Canagliflozin 100 mg Type=1 unit=mg number=100 form=tablet route=oral use. Tablet is taken once without food during 1 of 3 treatment periods.,Canagliflozin 300 mg Type=1 unit=mg number=300 form=tablet route=oral use. Tablet is taken once without food during 1 of 3 treatment periods.,Canagliflozin 50 mg Type=1 unit=mg number=50 form=tablet route=oral use.Tablet is taken once without food during 1 of 3 treatment periods.
  Interventions: Drug: Canagliflozin, 50 mg; Drug: Canagliflozin, 300 mg; Drug: Canagliflozin, 100 mg

INTERVENTIONS:
Drug: Canagliflozin, 50 mg — Type=1, unit=mg, number=50, form=tablet, route=oral use.Tablet is taken once without food during 1 of 3 treatment periods.
Drug: Canagliflozin, 300 mg — Type=1, unit=mg, number=300, form=tablet, route=oral use. Tablet is taken once without food during 1 of 3 treatment periods.
Drug: Canagliflozin, 100 mg — Type=1, unit=mg, number=100, form=tablet, route=oral use. Tablet is taken once without food during 1 of 3 treatment periods.

SUMMARY:
The purpose of this study is to evaluate the effect of dose on the pharmacokinetics of canagliflozin in healthy volunteers.

DETAILED DESCRIPTION:
This is an open-label study where healthy volunteers will know the name and dose of assigned treatment and will be randomly assigned to take a single oral (by mouth) dose of canagliflozin sequentially in each of 3 treament periods where the dose in each treatment period will be different (referred to as a 3-period crossover study) to evaluate the pharmacokinetics (blood levels) of 3 dose levels of canagliflozin. Healthy volunteers will take a single oral tablet of canagliflozin 50 mg (Treatment A), 100 mg (Treatment B), and 300 mg (Treatment C) during the study; a different dose will be taken in each treatment period. Study drug will be taken in the a.m. on Day 1 of Treatment Periods 1, 2, and 3, with a 10- to 14-day washout period between Day 1 of each treatment period. Volunteers will fast (go without food) for at least 10 hours before and up to at least 4 hours after taking study drug.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers with a body mass index between 18 and 30 kg/m2 (inclusive) and body weight not less than 50 kg

Exclusion Criteria:

* History of or current medical illness deemed clinically significant by the Investigator (study physician)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of canagliflozin | For up to 12 days (4 days during treatment periods 1, 2, and 3)

SECONDARY OUTCOMES:
Adverse events | Up to approximately 42 days (includes up to 14 days between Treatment Periods 1 and 2 and up to 10 days after Day 4 of Treatment Period 3)
Clinical laboratory tests | Up to approximately 42 days
Physical examinations | Up to approximately 42 days
12-lead electrocardiograms (ECGs) | Up to approximately 42 days
Vital signs | Up to approximately 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Merksem, Belgium

REFERENCES:
- [Derived] Devineni D, Manitpisitkul P, Murphy J, Stieltjes H, Ariyawansa J, Di Prospero NA, Rothenberg P. Effect of food on the pharmacokinetics of canagliflozin, a sodium glucose co-transporter 2 inhibitor, and assessment of dose proportionality in healthy participants. Clin Pharmacol Drug Dev. 2015 Jul;4(4):279-86. doi: 10.1002/cpdd.151. Epub 2014 Dec 11. PMID 27136908